CLINICAL TRIAL: NCT01993537
Title: The Role of Vitamin D in the Pathophysiology of Chronic Failure: Insight in to Mechanisms of Action and Implications for Vitamin D Supplementation
Brief Title: The Role of Vitamin D in the Pathophysiology of Chronic Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Responsible Party: Principal Investigator, Haissam Haddad, Director Heart Failure Program, Medical Director Heart Transplant Program, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120585
Record Dates: First submitted 2013-10-04; First posted 2013-11-25 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Vitamin D Deficiency; Chronic Heart Failure
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sufficeint (No Intervention): In this arm the participants have a Vitamin D level of greater than 75 ng/ml. They will continue to be monitored throughout the study but will not receive any intervention.
- Mild Insufficiency (No Intervention): In this arm the participants have a Vitamin D level between 37.5 - 75 ng/ml. The participants will be monitored throughout the study but will receive no intervention.
- Severe Deficiency no treatment (No Intervention): In this arm the participants have a low Vitamin D level of less than 37.5 ng/ml. The participants will be monitored but will receive no intervention.
- Severe Deficiency - Treatment (Experimental): In this arm the participants will be treated with Vitamin D. The participants will be prescribed a dose of 1000 IU a day (1 pill a day). At 6 weeks the dosage will increase to 2000 IU a day (2 pills a day).
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D
  Arms: Severe Deficiency - Treatment

SUMMARY:
Patients will undergo at baseline and regular intervals:

* clinically indicated bloodwork/urine and echocardiogram testing
* biomarker studies

Upon enrolment in the study patients will be divided into 4 groups normal, mildly deficient and severely deficient. Normal and mild vitamin D levels will receive no treatment while severe Vitamin D deficiency will be randomized (50/50) to receive no treatment or vitamin D treatment. They will be seen in the heart failure clinic every 6 months. The patients will be followed for 26 months.

DETAILED DESCRIPTION:
The inclusion criteria for the study is:

* an EF ≤40% within the last 12 months before recruitment
* established diagnosis of heart failure
* >18 years of age
* patients will vitamin d levels of sufficient, mild deficiency and severe deficiency

The exclusion criteria is:

* hypercalcemia
* known hypersensitivity to Vitamin D
* patient unwilling to comply with study requirements
* any other disease other than heart failure that can alter the patients quality of life over a period of 6 months
* women of child bearing potential
* a patient currently taking vitamin d
* severe renal impairment estimated glomerular filtration rate (eGFR) <30

ELIGIBILITY:
Inclusion Criteria:

* an ejection fraction (EF) ≤40% within the last 12 months before recruitment
* established diagnosis of heart failure
* >18 years of age
* patients with Vitamin D levels of sufficient, mild deficiency and severe deficiency

Exclusion Criteria:

* hypercalcemia
* known hypersensitivity to Vitamin D
* patient unwilling to comply with study requirements
* any other disease other than heart failure that can alter the patients quality of life over a period of 6 months
* women of child bearing potential
* a patient currently taking vitamin d
* severe renal impairment eGFR <30

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2013-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
prevalence of Vitamin D deficiency amongst chronic heart failure patients at the University of Ottawa Heart Institute | up to 3 years
  The primary outcome for the study is to identify the prevalence of Vitamin D deficiency amongst chronic heart failure patients followed at the University of Ottawa Heart Institute. This will be done analyzing the Vitamin D blood levels at baseline.

SECONDARY OUTCOMES:
To demonstrate that Vitamin D deficiency is associated with poor outcome and that Vitamin D supplementation can be of clinical benefit | up to 3 years
  clinical endpoints of: hospitalizations for worsening congestive heart failure, death will be compared for severe Vitamin D deficient patients receiving Vitamin D supplementation vs severe Vitamin D deficient patients receiving no intervention

CONTACTS AND LOCATIONS:
Overall Officials: Haissam Haddad, Principal Investigator — The University of Ottawa Heart Insitute
Locations (1):
- The University of Ottawa Heart Institute, Ottawa, Ontario, Canada